CLINICAL TRIAL: NCT00604487
Title: Induction of Labor in Patients With Unfavorable Cervical Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Principal Investigator, elad mei-dan, Elad Mei-Dan, MD, Hillel Yaffe Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: inductionCTIL; no grant
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Unfavorable Cervix for Induction of Labor
Keywords: induction; cervix; balloon; Bishop
MeSH Terms: interventions — Insemination, Artificial, Heterologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Insertion of the Atad double balloon ripener device (100 ml NS in each balloon).
  Interventions: Device: ARD (Atad Ripener Device)
- 2 (Active Comparator): Insertion of the double balloon instillation device (100 ml NS in each balloon) and continuous extra-amniotic instillation of NS 50 Ml/hour
  Interventions: Device: AID (Atad double balloon Instillation Device)
- 3 (Active Comparator): Insertion of the folly catheter (40 ml NS in the balloon) and continuous extra-amniotic instillation of NS 50 Ml/hour
  Interventions: Device: folly catheter

INTERVENTIONS:
Device: ARD (Atad Ripener Device) — Atad double balloon ripener device
  Arms: 1
Device: AID (Atad double balloon Instillation Device) — Double balloon instillation device and continuous extra-amniotic instillation of NS 50 Ml/hour
  Arms: 2
Device: folly catheter — folly catheter (40 ml NS in the balloon) and continuous extra-amniotic instillation of NS 50 Ml/hour
  Arms: 3

SUMMARY:
Artificial ripening of the cervix and induction of labor remain as one of the therapeutic challenges in Obstetrics. The method widely used, the intravenous administration of Oxytocin, is associated with prolonged induction periods, a significant failure rate, and considerable patient discomfort. Therefore, over the years, a variety of locally applied pharmacological and physical ripening agents were evaluated. Currently, the commonly utilised local ripening agent is a Prostaglandin (PG) preparation. Although PG is being applied vaginally or extra-amniotically, systemic absorption of this agent is common, sometimes resulting in uterine hypertonicity, nausea and vomiting. In addition, both induction methods are associated with the initiation of uterine contractions, sometimes lasting for prolonged periods. Therefore a preferred induction method may be a mechanical one which will lead to cervical ripening without causing uterine contractions. Furthermore, there are additional potential advantages of mechanical methods compared to pharmacologic methods such as, ease of storage, low cost and less side effects. A folly catheter, inserted through the cervix, combined with continuous extra-amniotic NS instillation is being used for this purpose for many years. However this method although effective may cause uncomfortable traction of the balloon to the women's leg. Furthermore, dripping of saline through the cervix and vagina, occasionally occurs, may be annoying, and may be confused with rupture of membrane. We have recently introduced a newly developed balloon device (Atad Ripener Device), which was designed with one balloon located at the distal end of the device (the uterine balloon, U), while the other balloon is located 1.5 cm proximal to the first one (the cervicovaginal balloon, CV). Both balloons are expandable with Saline. The balloon inflated in the vagina provides the traction action and seals the cervix from saline leakage. Another balloon the AID (Atad double balloon Instillation Device) is identical to the ARD but has an additional long tip for instillation of normal to the extra-amniotic space. To the best of our knowledge, no comparison was performed between the use of the double balloon ripener device and folly catheter for induction of labor. Furthermore, there are no published data regarding the use of the double balloon instillation device (AID) combined with continuous extra-amniotic NS instillation. This study is designed to compare the efficacy, safety and side effects of mechanical methods of cervical ripening and labor induction by the double balloon device (ARD), the double balloon instillation device (AID) combined with continuous extra-amniotic instillation of normal saline and the folly catheter combined with continuous extra-amniotic normal saline instillation. The study aims at the accrual of 300 women (100 randomised in each arm).

ELIGIBILITY:
Inclusion Criteria:

* Patients 15 years of age or older.
* Diagnosed to be pregnant with an indication for induction of labor.
* Having a Bishop score of 4 points or less.
* Diagnosed as having a singleton pregnancy in a vertex presentation, with intact membranes, and no significant regular uterine contraction at gestational age of >28 weeks.
* Willingness to comply with the protocol for the duration of the study.
* Have signed an informed consent.

Exclusion Criteria:

* Any contraindication for a vaginal delivery (i.e. placenta previa, non vertex presentation).
* Ruptured membranes.
* Previous cesarean section or any uterine scar.
* Documented labor.
* Suspected fetal distress necessitating immediate intervention.
* Proven malignancy of the cervix.
* Active inflammatory or purulent condition of the lower genital tract.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2008-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To evaluate and compare the efficacy of the Atad Ripening Device (ARD), of the double balloon instillation device (AID) with concomitant continuous extra-amniotic NS instillation - 50 Ml/hour and of the folly catheter combined with continuous extra-a | 2 years

SECONDARY OUTCOMES:
To assess the safety of the induction methods. | 2 years
To assess the women's experience and satisfaction with the induction methods. | 2 years
To compare the different cervical scoring systems available for predicting a successful induction. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai Hallak, M.D., Principal Investigator — Department of Obstetrics & Gynecology, Hillel Yaffe Medical Center, Hadera
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264
- [Derived] Anabusi S, Mei-Dan E, Hallak M, Walfisch A. Mechanical labor induction in the obese population: a secondary analysis of a prospective randomized trial. Arch Gynecol Obstet. 2016 Jan;293(1):75-80. doi: 10.1007/s00404-015-3765-3. Epub 2015 Jun 9. PMID 26054823
- [Derived] Walfisch A, Mei-Dan E, Hallak M. Trans-cervical double balloon catheter with and without extra-amniotic saline infusion for cervical ripening: a prospective quasi-randomized trial. J Matern Fetal Neonatal Med. 2015 May;28(7):848-53. doi: 10.3109/14767058.2014.935328. Epub 2014 Jul 11. PMID 24939630
- [Derived] Mei-Dan E, Walfisch A, Valencia C, Hallak M. Making cervical ripening EASI: a prospective controlled comparison of single versus double balloon catheters. J Matern Fetal Neonatal Med. 2014 Nov;27(17):1765-70. doi: 10.3109/14767058.2013.879704. Epub 2014 Feb 3. PMID 24397244